CLINICAL TRIAL: NCT03968003
Title: Impact of Dietary Fiber as Prebiotics on Intestinal Microbiota in Obese Thai Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 639/2017
Record Dates: First submitted 2019-05-09; First posted 2019-05-30 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2020-07

CONDITIONS: Obesity
Keywords: Prebiotics; Intestinal Microbiota
MeSH Terms: conditions — Obesity | interventions — Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: 165 participants Children, age 7 to 15 years with Body mass index (BMI) ≥ median + 2 Standard deviation(SD) will be randomized into one of the three arms of 55 participants per group. Group A (intervention group) will receive inulin 10 g. Group B will receive placebo of isocaloric maltodextrin. Group C will receive dietary fiber advice aimed to match the recommended fiber intake for age.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inulin (Experimental): Group A consumed 10 g of inulin extracted from Thai Jerusalem artichoke by our patent technique (Patent no. 15858) administered once daily before dinner.
  Interventions: Dietary Supplement: Inulin
- Maltodextrin (Placebo Comparator): Group B received isocaloric maltodextrin.
  Interventions: Dietary Supplement: Inulin
- Dietary fiber (Active Comparator): Group C will receive dietary fiber advice aimed to match age-appropriate intake recommendations.
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: Inulin — The intervention group (group A) consumed 10 g of inulin extracted from Thai Jerusalem artichoke by our patent technique (Patent no. 15858) administered once daily before dinner. The placebo group (group B) received isocaloric maltodextrin, while the dietary fiber advice group (group C) received guidance based on age-appropriate intake recommendations.
  Other Names: Maltodextrin

SUMMARY:
This study evaluates the changes of gut microbiota composition and diversity, gut-muscle axis, body weight, body fat, children eating behaviours, SCFAs, plasma amino acids, satiety hormones (Peptide-YY(PYY) and glucagon-like peptide 1(GLP-1)), Inflammatory cytokines (Interleukin-1β(IL-1β), Tumor necrosis factor-α (TNF-α) and Interleukin-6(IL-6)) after 6-month studied period in obese Thai children.165 participants Children, age 7 to 15 years with Body mass index (BMI) ≥ median + 2 standard deviation(SD) will be randomized into one of the three arms of 55 participants per group.Group A (intervention group) will receive inulin 10 g.Group B will receive placebo of isocaloric maltodextrin. Group C will receive dietary fiber advice aimed to match the recommended fiber intake for age.

DETAILED DESCRIPTION:
The prevalence of childhood obesity is increasing worldwide. The prevalence of overweight and obesity in children and adolescents has risen dramatically from 4% to 18% in 40 years.

Cause of obesity is gene-environment interactions. Recent evidence suggests that the gut microbiota is involved in energy regulation as well as inflammation Definition of obesity for children and teens is defined as a BMI at or above median +2 standard deviation(SD) of the same age and sex from World Health Organization (WHO) reference Management of childhood obesity are therapeutic lifestyle change by changing dietary habits and the physical activity level. Consumption of prebiotics, which are non-digestible polysaccharides that utilized by gut microorganisms then microbial shifts in response to prebiotic intake change in Bifidobacterium and lead to decreased body weight and adiposity. The microbial metabolite short-chain fatty acids (SCFAs) are likely to have impacts on various aspects of host physiology and then may decrease in body weight and adiposity.

The mechanism of inflammation in obesity, Lipopolysaccharides (LPS) which derived from the outer cell membrane of Gram-negative bacteria are the trigger factor of inflammation.LPS cross the gastrointestinal mucosa, then they reach the systemic circulation and trigger innate immune response activate the maturation of IL-1β. Circulating LPS levels were associated with elevated TNF-α and IL-6 concentrations in adipocytes.

Inulin-type fructans are non-digestible, fully soluble, and fermentable food ingredients with known prebiotic properties, which are found naturally in chicory root and Jerusalem artichoke, a plant grown in Thailand, that are fermented in the colon to produce SCFA. Bifidobacteria are preferentially stimulated to grow, by increasing the number of health-promoting bacteria and reducing the number of potentially harmful species.

There was only one study about the effect of prebiotics on composition of the intestinal microbiota in children with overweight or obesity. The study performed a randomized controlled trial to study children, 7-12 years old, with overweight or obesity. Participants were randomly assigned to groups given either oligofructose-enriched inulin (OI; 8 g/day; n = 22) or maltodextrin placebo (isocaloric dose, controls; n = 20) once daily for 16 weeks. Fecal samples were collected at baseline and 16 weeks and the composition of the microbiota was analyzed by 16S ribosomal ribonucleic acid (rRNA) sequencing and qPCR. The primary outcome was change in percent body fat from baseline to 16 weeks. After 16 weeks, quantitative polymerase chain reaction(qPCR) showed a significant increase in Bifidobacterium spp. in the OI group compared with controls. 16S rRNA sequencing revealed significant increases in species of the genus Bifidobacterium and decreases in Bacteroides vulgatus within the group who consumed OI.children who consumed OI had significant decreases in body weight z-score (decrease of 3.1%), percent body fat (decrease of 2.4%), percent trunk fat (decrease of 3.8%), interleukin 6 from baseline (decrease of 15%) compared with children given placebo.

ELIGIBILITY:
Inclusion Criteria:

* Children, age 7 to 15 years
* Body mass index (BMI) ≥ median + 2 Standard deviation (SD)

Exclusion Criteria:

* Underlying disease of syndromic obesity and monogenic obesity
* Endocrine causes of obesity (e.g. hypothyroidism, growth hormone deficiency)
* Use of drugs that influence appetite or body weight (e.g. corticosteroids)
* Attending other concurrent weight reduction programs

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in gut microbiota (16S rRNA sequencing) at 3 and 6 months | From the enrollment to 3 months and the end of intervention at 6 months.
  Gut microbial taxa, including Bifidobacterium, Blautia, Megasphaera, and several butyrate-producing bacteria, including Agathobacter, Eubacterium coprostanoligenes, and Subdoligranulum are being assessed.

SECONDARY OUTCOMES:
Change from baseline in Body mass index (BMI) at 1,2,3,4,5 and 6 months | From the enrollment to monthly visit and the end of intervention at 6 months.
  BMI was calculated as weight in kilograms divided by the square of height in meters (kg/m^2)
Change from baseline in fat mass index (FMI) at 6 months | From the enrollment to 3 months and the end of intervention at 6 months.
  FMI was calculated as weight of fat mass in kilograms divided by the square of height in meters (kg/m^2)
Change from baseline in fecal short chain fatty acids (SCFAs) at 3 and 6 months | From the enrollment to 3 months and the end of intervention at 6 months.
  fecal acetate, propionate and butyrate analyzed by using High Performance Liquid Chromatography (HPLC)
Change from baseline in Inflammatory cytokines (ELISA method)(IL-1β, TNF-α and IL-6) at 6 months | From the enrollment to the end of intervention at 6 months.
  Inflammatory cytokine (ELISA methods) (IL-1β (pg/ml), TNF-α (pg/ml) and IL-6 (pg/ml))
Change from baseline in Children Eating Behaviors at 3 and 6 months | From the enrollment to 3 months and the end of intervention at 6 months.
  Children eating behavior questionnaires (CEBQs) is constructed to assess eight aspects of children's eating behavior. There are four subscales that measure food-approach behaviors (food responsiveness, enjoyment of food, emotional overeating, and desire to drink) and the remaining four subscales measure food-avoidant behaviors (satiety responsiveness, slowness in eating, emotional undereating, and food fussiness). Each subscale comprises 3-6 items rated on a five-point Likert scale (scores range from 1 = never to 5 = always).
Change from baseline in serum GLP-1 hormone at 6 months. | From enrollment to the end of intervention at 6 months
  Glucagon-like peptide 1 (GLP-1) is measured in unit expressed as ng/L.
Change from baseline in PYY hormone at 6 months | From enrollment to the end of intervention at 6 months.
  Peptide YY (PYY) is measured in unit expressed pg/mL.
Change from baseline in myokine (interleukin-15) at 6 months | From enrollment to the end of intervention at 6 months.
  Myokine (interleukin-15 (IL-15)) is analyzed by enzyme-linked immunosorbent assay (ELISA) expressed as pg/mL.
Change from baseline in creatinine/cystatin C ratio at 6 months | From enrollment to the end of intervention at 6 months.
  Serum creatinine is measured using an enzymatic method on the Alinity C analyzers (mg/dL), and cystatin C assessed using particle-enhanced immunonephelometry using the BN Systems (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Chonnikant Visuthranukul, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Informed Consent Form will be available to share with other researchers.
Supporting Information: ICF
Time Frame: Data will become available in 2022 and will share for 1 year.
Access Criteria: Data will be made available upon request pending application and approval.

REFERENCES:
- [Result] Visuthranukul C, Leelahavanichkul A, Tepaamorndech S, Chamni S, Mekangkul E, Chomtho S. Inulin supplementation exhibits increased muscle mass via gut-muscle axis in children with obesity: double evidence from clinical and in vitro studies. Sci Rep. 2024 May 16;14(1):11181. doi: 10.1038/s41598-024-61781-1. PMID 38755201
- [Result] Visuthranukul C, Sriswasdi S, Tepaamorndech S, Chamni S, Leelahavanichkul A, Joyjinda Y, Aksornkitti V, Chomtho S. Enhancing gut microbiota and microbial function with inulin supplementation in children with obesity. Int J Obes (Lond). 2024 Dec;48(12):1696-1704. doi: 10.1038/s41366-024-01590-8. Epub 2024 Jul 20. PMID 39033197
- [Result] Visuthranukul C, Sriswasdi S, Tepaamorndech S, Joyjinda Y, Saengpanit P, Kwanbunbumpen T, Panichsillaphakit E, Uaariyapanichkul J, Chomtho S. Association of Human Intestinal Microbiota with Lifestyle Activity, Adiposity, and Metabolic Profiles in Thai Children with Obesity. J Nutr Metab. 2022 May 20;2022:3029582. doi: 10.1155/2022/3029582. eCollection 2022. PMID 35637874
- [Result] Visuthranukul C, Chamni S, Kwanbunbumpen T, Saengpanit P, Chongpison Y, Tepaamorndech S, Panichsillaphakit E, Uaariyapanichkul J, Nonpat N, Chomtho S. Effects of inulin supplementation on body composition and metabolic outcomes in children with obesity. Sci Rep. 2022 Jul 29;12(1):13014. doi: 10.1038/s41598-022-17220-0. PMID 35906473
- [Result] Visuthranukul C, Kwanbunbumpen T, Chongpison Y, Chamni S, Panichsillaphakit E, Uaariyapanichkul J, Maholarnkij S, Chomtho S. The Impact of Dietary Fiber as a Prebiotic on Inflammation in Children with Obesity. Foods. 2022 Sep 15;11(18):2856. doi: 10.3390/foods11182856. PMID 36140983
- [Result] Panichsillaphakit E, Chongpison Y, Saengpanit P, Kwanbunbumpen T, Uaariyapanichkul J, Chomtho S, Pancharoen C, Visuthranukul C. Children's Eating Behavior Questionnaire Correlated with Body Compositions of Thai Children and Adolescents with Obesity: A Pilot Study. J Nutr Metab. 2021 Jan 15;2021:6496134. doi: 10.1155/2021/6496134. eCollection 2021. PMID 33510908
- [Result] Saengpanit P, Chomtho S, Sriswasdi S, Rodpan A, Joyjinda Y, Panichsillaphakit E, Uaariyapanichkul J, Tempark T, Bongsebandhu-phubhakdi C, Suteerojntrakool O, Visuthranukul C. Dietary fiber intake and its relationships with lipid profiles and gut microbiota in obese Thai children: a pilot study. J Med Assoc Thai . 2019;102:1282-8.
- [Derived] Andriyas T, Sriswasdi S, Tansawat R, Uaariyapanichkul J, Chomtho S, Visuthranukul C. Inulin supplementation modulates gut microbiota derived metabolites related to brain function in children with obesity. Sci Rep. 2025 Oct 7;15(1):34843. doi: 10.1038/s41598-025-21079-2. PMID 41057493